# **Study Title:**

Demonstration Study of the Effect of Transcranial Direct Current Stimulation (tDCS) for Patients with Depression in Clinical Fields

NCT No.: NCT05539131

Date of Creation: March 23, 2023

# Study Protocol with Statistical Analysis Plan (SAP)

**Study Title:** Demonstration Study of the Effect of Transcranial Direct Current Stimulation (tDCS) for Patients with Depression in Clinical Fields

# **Study Protocol**

### **Purpose**

- 1. Demonstrate the clinical effectiveness of transcranial direct current stimulation (tDCS) for patients with depression in real-world clinical settings.
- 2. Optimize home-based electroceutical technologies for patient-centered applications.
- 3. Generate real-world data (RWD) and evidence (RWE) to support the adoption of tDCS in clinical practice.

# Design

#### 1. Overview:

- o Randomized, double-blinded, multi-site clinical study.
- Participants: 198 adults aged 19–65 with mild to moderate major depressive disorder (MDD).
- Duration: 6 weeks of home-based self-applied tDCS.

#### 2. Device:

o MINDD STIM+ (YMS-201B+/201BS+), an FDA-approved tDCS device.

# 3. Randomization:

- o Group A: Active tDCS for 6 weeks.
- Group B: Active tDCS for 3 weeks followed by 3 weeks of sham stimulation.

## 4. Primary Outcome Measures:

 Changes in BDI-II (Beck Depression Inventory-II) and MADRS (Montgomery-Åsberg Depression Rating Scale) scores from baseline (V1) to week 6 (V3).

## 5. Secondary Outcome Measures:

- HAM-A (Hamilton Anxiety Rating Scale) for anxiety.
- o DSST (Digit Symbol Substitution Test) for cognitive function.
- CESD-R for daily depressive symptom assessment.
- o qEEG (quantitative EEG) and HRV (heart rate variability).

## **Participant Criteria**

#### Inclusion:

- o Age 19–65, mild to moderate MDD diagnosis.
- o Informed consent capability.

#### • Exclusion:

- PTSD, psychotic MDD, severe suicidal risk, cranial implants, major cardiovascular or neurological issues.
- o Prior tDCS use or participation in clinical trials within 30 days.

# **Statistical Analysis Plan (SAP)**

#### **General Overview**

The statistical analysis will evaluate both primary and secondary outcomes based on intention-to-treat (ITT) and per-protocol (PP) populations.

# **Primary Statistical Methods**

## 1. Primary Analysis:

- Dependent Variables: Changes in BDI-II and MADRS scores from baseline to week 6.
- Methodology:
  - Independent t-tests to compare mean score changes between groups.
  - Mixed-effects models to adjust for repeated measures and site-level variation.

## 2. Secondary Analysis:

 Evaluate changes in HAM-A, DSST, and CESD-R scores over time using regression analysis.

# **Adjustments for Multiple Comparisons**

To control for Type I error:

• Bonferroni correction for the analysis of multiple secondary outcomes.

# **Handling Missing Data**

- Multiple imputation for missing data assuming data are missing at random (MAR).
- Sensitivity analysis to validate robustness.

# **Validation of Assumptions**

- 1. Normality: Shapiro-Wilk test for residuals.
- 2. Homogeneity of Variance: Levene's test.
- 3. **Sphericity (if repeated measures):** Mauchly's test.

# **Safety Analysis**

- Descriptive statistics for adverse events (AEs) and serious adverse events (SAEs).
- AE rates compared using Fisher's exact test or chi-square test.